CLINICAL TRIAL: NCT06231186
Title: Isotoxic High Dose (iHD) Fractionated Stereotactic Radiation Therapy (fSRT) for Intact Brain Metastases : a Feasibility Study
Brief Title: a Feasibility Study of iHD-SRT for BM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, JIAYI CHEN, Prof, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024（006）
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Brain Metastases, Adult; Stereotactic Radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iHD-SRT (Experimental): isotoxic high dose SRT
  Interventions: Radiation: iHD-SRT

INTERVENTIONS:
Radiation: iHD-SRT — received isotoxic individualized fSRT, with BED 10>50Gy and <100Gy, and strict OAR limits

SUMMARY:
Brain metastasis is the most challenging disease in the field of tumor treatment, with a median overall survival of only 1-2 months for untreated patients. Stereotactic radiotherapy (SRT) has the advantages of precise positioning, relatively concentrated dosage, shorter course, and lower toxicity. Several studies could effectively protect cognitive function and achieve better tumor control rate. Currently, it has gradually replaced WBRT as standard local treatment choice for brain metastases. SRT includes Stereotactic Radiosurgery (SRS) and Fractional Stereotactic Radiotherapy (fSRT). With the continuous updating of domestic radiation therapy equipment, the use of high-resolution multi leaf gratings enables the accuracy of fSRT based on linear accelerators to reach 0.5mm or even lower levels, and has gradually become one of the main choices for local treatment of a limited number of patients with brain metastases.

However, there is currently no prospective randomized controlled study data analyzing the clinical benefits of different segmentation and dosages of SRT. In retrospective data comparing different segmentation schemes, researchers found that higher BED was associated with better local control. However, the ASTRO guidelines recommend relatively conservative doses for SRT of brain metastases, especially as the lesion volume increases, and the recommended dose of BED10 for SRT was only 48 Gy (30 Gy/5 Fx). This is based on the consideration that higher radiation exposure will bring a higher risk of radiation-induced brain necrosis. However, with the continuous updates of SRT treatment equipment and technology, existing technologies can achieve higher dose coverage for more brain metastases while meeting the normal tissue limit. Therefore, this study conducted a prospective intervention study to explore the feasibility and safety of optimizing SRT dosage based on normal tissue tolerance for the treatment of brain metastases, in order to further improve the therapeutic effect of intracranial lesions with brain metastases.

This study is designed as a single arm open prospective study, assuming that under this treatment regimen, the proportion of patients with lesion prescription dose BED10>50 Gy is 90%, and the incidence of radiation-induced brain necrosis within 1 year is 8.5%. The planned enrollment period is 2 years and follow-up period is 1 year. A total of 35 people need to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to participate the research and sign the consent form
* ECOG PS 0-2
* The primary or metastatic lesion was confirmed by pathological histology as a malignant tumor
* Head MRI diagnosis of brain metastasis with measurable lesions and technically feasible SRT (no more than 15 in number and 20cc in volume)
* Estimated survival time ≥ 3 months

Exclusion Criteria:

* Diffuse brain metastases, or combined with meningeal metastases, or technically difficult to perform SRT
* With severe internal medicine complications or absolute contraindications for radiotherapy
* other sufficient reasons to be unqualified, such as potential non-compliance with the clinical protocol, etc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
proportion of patients receiving BED 10 >50 Gy | through treatment completion, an average of 1 month
  proportion of patients receiving BED 10 >50 Gy
the incidence of radiation-induced brain necrosis | 1 year
  The incidence of radiation-induced brain necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Chen, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided